CLINICAL TRIAL: NCT03487276
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Phase II Study to Determine Efficacy and Safety of IFX-1 in Subjects With Moderate to Severe Hidradenitis Suppurativa
Brief Title: Efficacy and Safety Study of IFX-1 in Patients With Moderate to Severe Hidradenitis Suppurativa (HS)
Acronym: SHINE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: InflaRx GmbH (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IFX-1-P2.4
Record Dates: First submitted 2018-02-27; First posted 2018-04-04 (Actual); Results first posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Hidradenitis Suppurativa (HS)
Keywords: hidradenitis suppurativa; monoclonal antibody; complement factor C5a; IFX-1; hidradenitis Suppurativa Clinical Response; Inflammation; skin diseases
MeSH Terms: conditions — Hidradenitis Suppurativa; Inflammation; Skin Diseases | interventions — vilobelimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Cohort 2 (Experimental): Minimum Dose IFX-1 (400 mg Q4W)
  Interventions: Drug: IFX-1
- Cohort 3 (Experimental): Low dose IFX-1 (800 mg Q4W)
  Interventions: Drug: IFX-1
- Cohort 4 (Experimental): Medium Dose IFX-1 (800 mg Q2W)
  Interventions: Drug: IFX-1
- Cohort 5 (Experimental): High Dose IFX-1 (1200 mg Q2W)
  Interventions: Drug: IFX-1

INTERVENTIONS:
Drug: IFX-1 — Single IV infusions of IFX-1 diluted in sodium chloride.
  Other Names: CaCP29; Vilobelimab
  Arms: Cohort 2; Cohort 3; Cohort 4; Cohort 5
Drug: Placebo — Placebo
  Arms: Cohort 1

SUMMARY:
The purpose of this study is to determine whether IFX-1 is safe and effective in the treatment of moderate to severe hidradenitis suppurativa.

DETAILED DESCRIPTION:
Hidradenitis suppurativa (HS) is a chronic devastating skin disorder affecting areas rich in apocrine glands. HS is diagnosed by its clinical features and its chronicity. It is recognized by the presence of recurrent, painful, deep-seated, rounded nodules usually ending in abscesses and sinus tracts with suppuration and hypertrophic scarring. As complement C5a is involved in the underlying acute inflammatory responses, this study is set up based on the hypothesis that IFX-1 might be able to block C5a induced pro-inflammatory effects such as neutrophil activation and cytokine generation, potentially contributing to the local skin inflammation and tissue damage.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ≥ 18 years of age
* Written informed consent obtained from subject
* Diagnosis of HS for at least 1 year
* Moderate or severe HS, as indicated by HS lesions in at least 2 distinct areas, 1 of which must be at least Hurley Stage II or Stage III
* Inadequate response to at least 3 months of oral antibiotics, or intolerance to antibiotics
* Total abscess and inflammatory nodule (AN) count of ≥ 3

Exclusion Criteria:

* Prior treatment with adalimumab or another biologic product during the 24 weeks before Screening
* Subjects on permitted oral antibiotic treatment for HS (doxycycline or minocycline only) who have not been on a stable dose during the 28 days before Screening
* Subject received systemic non-biologic therapy for HS with potential therapeutic impact for HS during the 28 days before Screening (other than permitted oral antibiotics)
* Prior treatment with any of the following medications during the 28 days before Screening:

  * Any other systemic therapy for HS
  * Any iv anti-infective therapy
  * Phototherapy (ultraviolet B or psoralen and ultraviolet A)
* History of heart disease or malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2019-05-27 (Actual); Study Completion 2020-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Othmar Zenker, CMO, Study Director — InflaRx GmbH
Locations (37):
- United States (12):
  - InflaRX Investigational Site, Birmingham, Alabama
  - InflaRX Investigational Site, Fort Myers, Florida
  - InflaRX Investigational Site, Miami, Florida
  - InflaRX Investigational Site, Sandy Springs, Georgia
  - InflaRX Investigational Site, Dearborn, Michigan
  - InflaRX Investigational Site, Columbia, Missouri
  - InflaRx Investigational Site, Saint Joseph, Missouri
  - InflaRX Investigational Site, St Louis, Missouri
  - InflaRX Investigational Site, Chapel Hill, North Carolina
  - InflaRX Investigational Site, Cincinnati, Ohio
  - InflaRX Investigational Site, Hershey, Pennsylvania
  - InflaRx Investigational Site, Goodlettsville, Tennessee
- Bulgaria (2):
  - InflaRX Investigational Site, Sofia
  - InflaRX Investigational Site, Stara Zagora
- Canada (3):
  - InflaRX Investigational Site, St. John's, Newfoundland and Labrador
  - InflaRX Investigational Site, Peterborough, Ontario
  - InflaRX Investigational Site, Richmond Hill, Ontario
- Denmark (2):
  - InflaRX Investigational Site, Copenhagen
  - InflaRX Investigational Site, Roskilde
- France (6):
  - InflaRX Investigational Site, Nice, Alpes Maritimes
  - InflaRX Investigational Site, Bordeaux, Gironde
  - InflaRX Investigational Site, Toulouse, Haute Garonne
  - InflaRX Investigational Site, Antony, Hauts De Seine
  - InflaRX Investigational Site, Nantes, Loire Atlantique
  - InflaRX Investigational Site, Paris
- Germany (4):
  - InflaRX Investigational Site, Darmstadt, Hesse
  - InflaRX Investigational Site, Frankfurt am Main, Hesse
  - InflaRX Investigational Site, Bochum, North Rhine-Westphalia
  - InflaRX Investigational Site, Dessau, Saxony-Anhalt
- Greece (2):
  - InflaRX Investigational Site, Athens
  - InflaRX Investigational Site, Thessaloniki
- InflaRX Investigational Site, Rotterdam, Netherlands
- Poland (5):
  - InflaRX Investigational Site, Gdansk
  - InflaRX Investigational Site, Krakow
  - InflaRX Investigational Site, Kłodzko
  - InflaRX Investigational Site, Lodz
  - InflaRX Investigational Site, Wroclaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Giamarellos-Bourboulis EJ, Jemec GBE, Prens EP, Riedemann NC, Otto I, Weisman J, Pulka G, Nowicki RJ, Kantardjiev V, Pinter A, Thomsen SF, Berneman D, Kanni T, Alavi A, Breno B, Gooderham M, Stone M, Anadkat MJ, Katoulis A, Papakonstantis M, Becherel PA, Szepietowski JC, van der Zee HH, Zouboulis CC, Sayed CJ. Vilobelimab to improve clinical outcomes in moderate-to-severe hidradenitis suppurativa through an adjunctive effect on draining tunnels: results of the SHINE double-blind placebo-controlled randomized trial. Br J Dermatol. 2026 Jan 27;194(2):254-263. doi: 10.1093/bjd/ljaf398. PMID 41081529
- [Derived] Prens LM, Ardon CB, van Straalen KR, van der Zee HH, Seelen MAJ, Laman JD, Prens EP, Horvath B, Damman J. No Evident Systemic Terminal Complement Pathway Activation in Hidradenitis Suppurativa. J Invest Dermatol. 2021 Dec;141(12):2966-2969.e1. doi: 10.1016/j.jid.2021.03.037. Epub 2021 Jul 9. No abstract available. PMID 34252397

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of a Main and an Extension Period. In the Main Period 175 subjects were planned to be randomized to receive double-blind treatment with IMP or Placebo in 1 of 5 treatment cohorts in a ratio of 1:1:1:1:1. The Extension Period started after the Week 16 Visit. According to the assessed HiSCR response at Week 16, patients were distributed to two IFX-1 dosing regimens: Week 16 HiSCR responders to 800 mg Q4W and Week 16 HiSCR non-responders to 800 mg Q2W.
Period: Main Period (16 Weeks)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Started | 37 | 34 | 36 | 36 | 36
Completed | 34 | 30 | 32 | 30 | 31 (One patient completed the Main Period but was lost to follow-up afterwards and not treated in the Extension Period)
Not Completed | 3 | 4 | 4 | 6 | 5
Period: Extension Period (28 Weeks)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Started | 0 | 0 | 72 | 84 | 0
Number of Patients in Cohort 1 (Main Period) Crossed Over to Cohort 3 or 4 | 0 | 0 | 16 | 18 | 0
Number of Patients in Cohort 2 (Main Period) Crossed Over to Cohort 3 or 4 | 0 | 0 | 12 | 18 | 0
Number of Patients in Cohort 3 (Main Period) Crossed Over to Cohort 3 or 4 | 0 | 0 | 17 | 15 | 0
Number of Patients in Cohort 4 (Main Period) Crossed Over to Cohort 3 or 4 | 0 | 0 | 12 | 18 | 0
Number of Patients in Cohort 5 (Main Period) Crossed Over to Cohort 3 or 4 (One patient of Cohort 5 completed the Main Period as Non-Responder but was lost to follow-up afterwards and not treated in the Extension Period) | 0 | 0 | 15 | 16 | 0
Completed | 0 | 0 | 67 | 54 | 0
Not Completed | 0 | 0 | 5 | 30 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis performed for safety analysis set (SAS)
Groups:
- Cohort 2: Minimum Dose IFX-1
  IFX-1: Single IV infusions of IFX-1 diluted in sodium chloride.
- Cohort 3: Low dose IFX-1
  IFX-1: Single IV infusions of IFX-1 diluted in sodium chloride.
- Cohort 4: Medium Dose IFX-1
  IFX-1: Single IV infusions of IFX-1 diluted in sodium chloride.
- Cohort 5: High Dose IFX-1
  IFX-1: Single IV infusions of IFX-1 diluted in sodium chloride.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Total
Number analyzed (Participants) | 36 | 34 | 35 | 36 | 36 | 177
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 35 | 33 | 35 | 36 | 35 | 174
  >=65 years | 1 | 1 | 0 | 0 | 1 | 3
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34.5 [27.0 to 42.5] | 39.0 [33.0 to 45.0] | 35.0 [25.0 to 46.0] | 37.0 [31.0 to 46.0] | 33.5 [27.5 to 41.0] | 36.0 [29.0 to 45.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 16 | 18 | 20 | 23 | 98
  Male | 15 | 18 | 17 | 16 | 13 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 1 | 4 | 7
  Not Hispanic or Latino | 36 | 33 | 34 | 35 | 32 | 170
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 4 | 4 | 4 | 17
  White | 33 | 31 | 29 | 32 | 27 | 152
  More than one race | 0 | 0 | 1 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 3 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  Greece | 9 | 5 | 9 | 10 | 14 | 47
  Canada | 1 | 0 | 2 | 4 | 1 | 8
  Netherlands | 2 | 0 | 1 | 1 | 2 | 6
  United States | 4 | 7 | 8 | 7 | 7 | 33
  Denmark | 2 | 2 | 1 | 0 | 0 | 5
  Poland | 11 | 9 | 4 | 8 | 6 | 38
  Bulgaria | 2 | 4 | 2 | 1 | 0 | 9
  France | 4 | 3 | 5 | 3 | 4 | 19
  Germany | 1 | 4 | 3 | 2 | 2 | 12
Baseline AN (total abscess and inflammatory nodule) count [Median (Inter-Quartile Range); unit: lesions] | 9.5 [5.0 to 15.0] | 9.0 [6.0 to 15.0] | 8.0 [7.0 to 17.0] | 10.0 [6.0 to 16.0] | 12.5 [5.5 to 15.5] | 9.0 [6.0 to 16.0]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Hidradenitis Suppurativa Clinical Response (HiSCR) Determined at Week 16
Description: The primary efficacy endpoint of the percentage of patients with HiSCR at Week 16 was analyzed using the multiple comparisons procedure-modelling (MCP-Mod) procedure. The definition for response to treatment based on HiSCR relative to Baseline was: at least 50% reduction in abscesses and inflammatory nodule (AN) count (over all anatomical regions) with no increase in number of abscesses and in number of draining fistulas.
Time Frame: Week 16
Population: Analysis was performed on the full analysis set (FAS) population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 34 | 30 | 33 | 31 | 33
Participants
  HiSCR Responder | 16 | 12 | 17 | 12 | 15
  HiSCR Non-responder | 18 | 18 | 16 | 19 | 18

2. Secondary Outcome: Number of Patients With Hidradenitis Suppurativa Clinical Response (HiSCR) Determined at Week 12
Description: Endpoint of the percentage of patients with HiSCR at Week 12 was analyzed in the same way as the primary endpoint using the MCP-Mod procedure and the same definition of response.
Time Frame: Week 12
Population: Analysis was performed on the full analysis set (FAS) population. Only patients with non-missing assessment at Week 12 were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 34 | 31 | 33 | 32 | 32
Participants
  HiSCR Responder | 14 | 14 | 12 | 13 | 13
  HiSCR Non-responder | 20 | 17 | 21 | 19 | 19

3. Secondary Outcome: Number of Patients With Flares Relative to Day 1
Description: The number of patients with flares analyzed in terms of ≥ 25% increase in abscess and inflammatory nodule (AN) count among patients with a minimum increase of 2 in AN count compared to Day 1 was analyzed by descriptive statistics by time point.
Time Frame: From Day 1 until Day 309
Population: For the Main Period the full analysis set was used for the analysis and results of Week 16 are displayed.
  For the Extension Period the safety analysis set was used for the analysis and results of week 44 are displayed.
  Only patients with non-missing assessment at the respective visit were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Main Period: Cohort 1: Placebo
  Placebo: Placebo
- Main Period: Cohort 2: Minimum Dose IFX-1 (400 mg Q4W)
  IFX-1: Single IV infusions of IFX-1 diluted in sodium chloride.
- Main Period: Cohort 3; Extension Period: Cohort 3: Low dose IFX-1 (800 mg Q4W)
  IFX-1: Single IV infusions of IFX-1 diluted in sodium chloride.
- Main Period: Cohort 4: Medium Dose IFX-1 (800 mg Q2W)
  IFX-1: Single IV infusions of IFX-1 diluted in sodium chloride.
- Main Period: Cohort 5: High Dose IFX-1 (1200 mg Q2W)
  IFX-1: Single IV infusions of IFX-1 diluted in sodium chloride.
- Extension Period: Cohort 4: Low dose IFX-1 (800 mg Q2W)
  IFX-1: Single IV infusions of IFX-1 diluted in sodium chloride.
Arm/Group | Main Period: Cohort 1 | Main Period: Cohort 2 | Main Period: Cohort 3 | Main Period: Cohort 4 | Main Period: Cohort 5 | Extension Period: Cohort 3 | Extension Period: Cohort 4
Number analyzed (Participants) | 34 | 30 | 32 | 30 | 32 | 67 | 52
Participants
  Patient with flares | 6 | 3 | 1 | 0 | 1 | 3 | 5
  Patient without flares | 28 | 27 | 31 | 30 | 31 | 64 | 47

4. Secondary Outcome: Absolute Change in Modified Sartorius Score (mSS) From Day 1.
Description: The absolute change from Day 1 will be analyzed by descriptive statistics by time point. The mSS is a summation of HS lesions based on a number of factors including anatomical region, number and type of lesions, distance between relevant lesions and lesions clearly separated by normal skin in each region measured as HS clinical parameters. The scale title for mSS is points. The mSS has a minimum value of 0 and no upper limit. The higher the score the more severe is the disease/worse is the outcome.
Time Frame: From Day 1 until Day 309
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Main Period: Cohort 1 | Main Period: Cohort 2 | Main Period: Cohort 3 | Main Period: Cohort 4 | Main Period: Cohort 5 | Extension Period: Cohort 3 | Extension Period: Cohort 4
Number analyzed (Participants) | 33 | 28 | 30 | 28 | 31 | 64 | 49
score on a scale | -16.4 (30.78) | -17.5 (48.43) | -29.4 (32.35) | -22.9 (52.00) | -35.2 (101.91) | -47.9 (70.87) | -27.5 (45.02)

5. Secondary Outcome: Absolute Change in Patient's Global Assessment of Skin Pain From Day 1.
Description: The absolute changes from baseline were analyzed by descriptive statistics by time point. The Numeric Rating Scale (NRS) was used to assess the worst skin pain due to HS. The scale title for the NRS is points. Ratings for this item range from a minimum of 0 points (no skin pain) to a maximum of 10 points (skin pain as bad as you can imagine). The higher the score the more severe the disease/worse is the outcome.
Time Frame: From Day 1 until Day 309
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Main Period: Cohort 1 | Main Period: Cohort 2 | Main Period: Cohort 3 | Main Period: Cohort 4 | Main Period: Cohort 5 | Extension Period: Cohort 3 | Extension Period: Cohort 4
Number analyzed (Participants) | 29 | 23 | 24 | 22 | 21 | 32 | 28
score on a scale | -1.2 (2.82) | -0.1 (2.68) | -0.7 (2.37) | -1.5 (2.92) | -1.8 (3.03) | -1.5 (2.94) | -1.3 (2.52)

6. Secondary Outcome: Percentage of Patients Achieving NRS30
Description: This is a segmented numeric version of the visual analog scale in which a respondent selects a whole number (0-10) that best reflects the intensity of their pain. The scale title for the NRS is points. The minimum score is 0 points (No skin pain), and the maximum score is 10 points (Skin pain as bad as you can imagine). The higher the score the more severe is the disease/worse is the outcome. The number of patients with at least 30% reduction and at least 1 point reduction from Day 1 in Patients Global Assessment of Skin Pain are displayed. The analysis is based on the worst skin pain the patients reported at the respective visits.
Time Frame: From Day 1 until Day 309
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Main Period: Cohort 1 | Main Period: Cohort 2 | Main Period: Cohort 3 | Main Period: Cohort 4 | Main Period: Cohort 5 | Extension Period: Cohort 3 | Extension Period: Cohort 4
Number analyzed (Participants) | 28 | 22 | 23 | 22 | 21 | 30 | 28
Participants | 7 | 6 | 5 | 9 | 8 | 12 | 10

7. Secondary Outcome: Percentage of Patients Achieving NRS50.
Description: This is a segmented numeric version of the visual analog scale in which a respondent selects a whole number (0-10) that best reflects the intensity of their pain. The scale title for NRS is points. The minimum score is 0 points (No skin pain), and the maximum score is 10 points (Skin pain as bad as you can imagine). The higher the score the more severe is the disease/worse is the outcome. The number of patients with at least 50% reduction and at least 1 point reduction from Day 1 in Patients Global Assessment of Skin Pain are displayed. The analysis is based on the worst skin pain the patients reported at the respective visits.
Time Frame: From Day 1 until Day 309
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Main Period: Cohort 1 | Main Period: Cohort 2 | Main Period: Cohort 3 | Main Period: Cohort 4 | Main Period: Cohort 5 | Extension Period: Cohort 3 | Extension Period: Cohort 4
Number analyzed (Participants) | 28 | 22 | 23 | 22 | 21 | 30 | 28
Participants | 6 | 3 | 2 | 7 | 5 | 7 | 5

8. Secondary Outcome: Absolute Change in Dermatology Life Quality Index (DLQI) Score From Day 1.
Description: The changes from Day 1 will be analyzed by descriptive statistics by time point. A score is documented for each of the 10 DLQI items, ranging from 0 to 3 for each item. The scale title for DLQI is points. The total score is the sum of the responses to all 10 DLQI items, ranging from the minimum of 0 points to the maximum of 30 points. A higher score corresponds to worse health related quality of life/outcome.
Time Frame: From Day 1 until Day 309
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Main Period: Cohort 1 | Main Period: Cohort 2 | Main Period: Cohort 3 | Main Period: Cohort 4 | Main Period: Cohort 5 | Extension Period: Cohort 3 | Extension Period: Cohort 4
Number analyzed (Participants) | 32 | 30 | 30 | 28 | 32 | 59 | 48
score on a scale | -1.5 (6.11) | 0.6 (6.39) | -2.6 (7.19) | -5.0 (5.90) | -2.4 (5.24) | -1.5 (7.18) | -2.0 (6.52)

9. Secondary Outcome: Safety Parameters (Adverse Events) Will be Assessed.
Description: The number of patients with any treatment emergent adverse event (adverse events that started after first infusion of IMP) was analyzed by time point.
Time Frame: From Day 1 until Day 309
Population: For the Main Period the safety analysis set was used for the analysis and results of Week 16 are displayed.
  For the Extension Period the safety analysis set was used for the analysis and results of week 44 are displayed.
  Only patients with non-missing assessment at the respective visit were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Period: Cohort 1 | Main Period: Cohort 2 | Main Period: Cohort 3 | Main Period: Cohort 4 | Main Period: Cohort 5 | Extension Period: Cohort 3 | Extension Period: Cohort 4
Number analyzed (Participants) | 36 | 34 | 35 | 36 | 36 | 72 | 84
Participants | 26 | 26 | 21 | 24 | 22 | 39 | 49

ADVERSE EVENTS:
Time Frame: The observation period for Adverse Events (AEs) will start with confirmation of signed informed consent at Screening and ends at the Follow-up visit at Week 44.
Description: The safety data were analyzed separately for the Main Period and the Extension Period. AEs assessed up to and including Week 16 Visit were attributed to the Main Period. All safety data assessed after IFX-1 infusion at Week 16 were attributed to the Extension Period. Analysis were performed in the safety analysis set consisting of 177 patients. Of the 179 randomized patients, only 177 received treatment with IMP as 2 patients withdrew from the study before they were treated.
Groups:
- Extension Period: Cohort 4: Medium Dose IFX-1 (800 mg Q2W)
  IFX-1: Single IV infusions of IFX-1 diluted in sodium chloride.
Arm/Group | Main Period: Cohort 1 | Main Period: Cohort 2 | Main Period: Cohort 3 | Main Period: Cohort 4 | Main Period: Cohort 5 | Extension Period: Cohort 3 | Extension Period: Cohort 4
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/34 | 0/35 | 0/36 | 0/36 | 0/72 | 0/84
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/34 | 1/35 | 2/36 | 3/36 | 2/72 | 3/84
Other Adverse Events (participants affected / at risk) | 26/36 | 26/34 | 21/35 | 24/36 | 22/36 | 34/72 | 49/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Main Period: Cohort 1 (N=36) | Main Period: Cohort 2 (N=34) | Main Period: Cohort 3 (N=35) | Main Period: Cohort 4 (N=36) | Main Period: Cohort 5 (N=36) | Extension Period: Cohort 3 (N=72) | Extension Period: Cohort 4 (N=84)
Abscess bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholangitis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Main Period: Cohort 1 (N=36) | Main Period: Cohort 2 (N=34) | Main Period: Cohort 3 (N=35) | Main Period: Cohort 4 (N=36) | Main Period: Cohort 5 (N=36) | Extension Period: Cohort 3 (N=72) | Extension Period: Cohort 4 (N=84)
Nasopharyngitis (Infections and infestations) | 6 | 4 | 6 | 4 | 3 | 4 | 8
Influenza (Infections and infestations) | 2 | 0 | 0 | 0 | 3 | 2 | 2
Pharyngitis (Infections and infestations) | 2 | 1 | 1 | 0 | 1 | 2 | 2
Sinusitis (Infections and infestations) | 0 | 0 | 2 | 1 | 1 | 1 | 0
Abscess (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 1 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Immune system disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 5 | 4 | 2 | 7 | 6 | 8 | 10
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 0 | 0 | 1 | 1
Fatigue (General disorders) | 2 | 0 | 3 | 2 | 3 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 2 | 3 | 1 | 2 | 2
Nausea (Gastrointestinal disorders) | 2 | 2 | 1 | 1 | 2 | 0 | 2
Viral upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 3
Pyrexia (General disorders) | 1 | 2 | 0 | 0 | 2 | 2 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 6 | 4 | 0 | 4 | 5 | 4 | 6
Syncope (Nervous system disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 1
International normalised ratio increased (Investigations) | 2 | 0 | 0 | 0 | 2 | 1 | 3
Foot fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 4
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 0 | 1 | 1 | 4
Hypertension (Vascular disorders) | 0 | 0 | 0 | 2 | 1 | 2 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-16): https://cdn.clinicaltrials.gov/large-docs/76/NCT03487276/Prot_SAP_000.pdf